CLINICAL TRIAL: NCT03773146
Title: A Randomized Controlled Trial of Varying Airtime Incentive Structure to Improve Interactive Voice Response (IVR) Survey Performance in Bangladesh and Uganda
Brief Title: Use of Airtime Structure to Improve Interactive Voice Response Surveys in Bangladesh and Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Makerere University (Other); Institute of Epidemiology, Disease Control and Research (Other); The Bloomberg Family Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00007318-2
Record Dates: First submitted 2018-12-05; First posted 2018-12-12 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2018-12

CONDITIONS: Surveys and Questionnaires; Noncommunicable Diseases
Keywords: mobile phone surveys; interactive voice response; incentive
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of three airtime incentive structures: 1) no incentive; 2) a fixed 1X incentive for all participants who completed the noncommunicable disease risk factor survey; or 3) a lottery incentive (10-20 times larger than the fixed incentive) given to 1 out of every 20 participants who completed the same survey.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No airtime incentive was given for completing the survey
- 1X Incentive (Experimental): 1X Airtime Incentive
  Interventions: Other: 1X Airtime Incentive
- Lottery (Experimental): Lottery Airtime Incentive
  Interventions: Other: Lottery Airtime Incentive

INTERVENTIONS:
Other: 1X Airtime Incentive — An incentive given in the form of airtime
  Arms: 1X Incentive
Other: Lottery Airtime Incentive — An incentive given in the form of airtime
  Arms: Lottery

SUMMARY:
This study evaluates the effect of three different airtime incentive structures on interactive voice response (IVR) survey cooperation, response, refusal and contact rates, as compared to a control group, in Bangladesh and Uganda.

DETAILED DESCRIPTION:
Using random digit dialing (RDD) sampling technologies, participants were randomized to one of three airtime incentive structures contingent on them completing the noncommunicable disease risk factor survey. This mobile phone survey was sent as an interactive voice response (IVR). In IVR surveys, participants use their touch tone key pad to answer pre-recorded questions. (i.e. if you are male, press 1; if you are female, press 2). This study is being conducted in both Bangladesh and Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone
* Greater or equal to 18 years of age
* In Bangladesh, conversant in either English or Bangla language. In Uganda, conversant in either Luo, Runyakitara, Luganda or English languages.

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4550 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Cooperation Rate #1 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, cooperation rate is defined as I/(I+P+R) where I is complete interviews, P is partial interviews, R is refusals and breakoffs
Response Rate #4 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, response rate is defined as (I+P)/ (I+P+R+eU) where I is complete interview, P is partial interview, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

SECONDARY OUTCOMES:
Refusal Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, refusal rate is defined as R/(I+P+R+eU) where R is refusals and breakoffs, I is complete interview, P is partial interview, and eU is the estimated eligible proportion of unknowns
Contact Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, contact rate is defined as (I+P+R)/ (I+P+R+eU) where I is complete interview, P is partial interview, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

CONTACTS AND LOCATIONS:
Overall Officials: Adnan A Hyder, PhD, MBBS, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; George W Pariyo, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (2):
- Institute of Epidemiology Disease Control and Research, Dhaka, Bangladesh
- Makerere University School of Public Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson DG, Pariyo GW, Wosu AC, Greenleaf AR, Ali J, Ahmed S, Labrique AB, Islam K, Masanja H, Rutebemberwa E, Hyder AA. Evaluation of Mechanisms to Improve Performance of Mobile Phone Surveys in Low- and Middle-Income Countries: Research Protocol. JMIR Res Protoc. 2017 May 5;6(5):e81. doi: 10.2196/resprot.7534. PMID 28476729
- [Background] Gibson DG, Pereira A, Farrenkopf BA, Labrique AB, Pariyo GW, Hyder AA. Mobile Phone Surveys for Collecting Population-Level Estimates in Low- and Middle-Income Countries: A Literature Review. J Med Internet Res. 2017 May 5;19(5):e139. doi: 10.2196/jmir.7428. PMID 28476725
- [Background] Gibson DG, Farrenkopf BA, Pereira A, Labrique AB, Pariyo GW. The Development of an Interactive Voice Response Survey for Noncommunicable Disease Risk Factor Estimation: Technical Assessment and Cognitive Testing. J Med Internet Res. 2017 May 5;19(5):e112. doi: 10.2196/jmir.7340. PMID 28476724
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722
- [Derived] Gibson DG, Kibria GMA, Pariyo GW, Ahmed S, Ali J, Labrique AB, Khan IA, Rutebemberwa E, Flora MS, Hyder AA. Promised and Lottery Airtime Incentives to Improve Interactive Voice Response Survey Participation Among Adults in Bangladesh and Uganda: Randomized Controlled Trial. J Med Internet Res. 2022 May 9;24(5):e36943. doi: 10.2196/36943. PMID 35532997